CLINICAL TRIAL: NCT06539104
Title: Scanning the Meiotic Spindle in Assisted Reproductive Techniques to Assess Oocyte Quality and Embryo Ploidy Evaluated by Artificial Intelligence (SMARTAI Study)
Brief Title: Aftificial Inteligence in Assisted Reproductive Techniques to Assess Oocyte Quality and Embryo Ploidy
Acronym: SMARTAI
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Czech Academy of Sciences (Other); Czech Technical University in Prague (Other); General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Jaromír Mašata, Leading doctor of the Center of Urogynecology and Pelvic Recontructive Surgery, Charles University, Czech Republic
Other Study IDs: NW24-08-00048
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Infertility; Infertility, Female; Infertility, Male; Infertility Unexplained
Keywords: infertility; humant oocyte; IVF; arteficial inteligence; Sperm count; meiotic spindle; time lapse
MeSH Terms: conditions — Infertility; Infertility, Female; Infertility, Male | interventions — Embryonic Development; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sperms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: arteficial inteligence evaluation of oocyte and embryo development — apply AI to find out the complex oocyte quality, embryo development, embryo ploidy and pregnancy success probability from the sequence of the data starting from the recording of the meiotic spindle in polarized light, through paternal factors up to the time lapse record of early embryo development.
  Other Names: Preimplantation Genetic Testing (PDT); Computer Assisted Sperm Analysis (CASA); DNA Sperm Fragmentation Index (DFI); Intracytoplasmatic Sperm Injection (ICSI)

SUMMARY:
The assisted reproduction success rate is affected by several factors including the age of the women, oocyte quality and maturation state, as well as sperm quality. Imaging of the meiotic spindle may be crucial for determining the oocyte maturation. Artificial intelligence (AI) will be applied to establish the complex oocyte quality, embryo ploidy and pregnancy success probability from the sequence of data, starting with the recording of the meiotic spindle in polarized light, through paternal factors up to the time lapse recording of early embryo development. This strategy should reduce the cost of fertility treatment thanks to increased efficiency in choosing the most promising candidates and reducing the need for costly laboratory analyses.

DETAILED DESCRIPTION:
One of the main strategies of infertility treatment is in vitro fertilization (IVF). The IVF success rate is affected by several key factors including the age of the women, oocyte quality and maturation state, as well as sperm quality. It has been suggested that the presence, position and retardance of the optically birefringent meiotic spindle (MS) are related to oocyte developmental competence, affecting the quality of fertilization and embryo development. Artificial intelligence (AI) will be applied to establish the complex oocyte quality, embryo ploidy and pregnancy success probability from the sequence of data, starting with the recording of the meiotic spindle in polarized light, through paternal factors up to the time lapse recording of early embryo development.

Synergic approaches will be used to increase the quality of embryos for implantation: image analysis and machine learning techniques will be applied to the oocyte microscopic images to perform the MS analysis fully automatically and to determine whether some other aspects of the oocyte appearance might correlate with the optimal timing and fertilization and pregnancy success, or genetic defects. An automatic method of embryo evaluation based on time-lapse videos after ICSI and MS imaging plus other scalar parameters (extracted features can be used as inputs for the downstream tasks, e.g. features extracted from oocytes and sperm can serve as additional inputs to the embryo classifier) will be used. This strategy should reduce the cost of fertility treatment thanks to increased efficiency in choosing the most promising candidates and reducing the need for costly laboratory analyses.

The analysis will be performed in cooperation with Czech Technical University and Institute of Physics Academy of Sciences of the Czech Republic who will create a software tool capable of predicting the probability of pregnancy and embryo ploidy status from oocyte images plus time-lapse video of a developing embryo after ICSI. It will be determined whether some other aspects of the oocyte appearance correlate with the fertilization and pregnancy success, or genetic defects.

Time lapse sequences of embryonic development and oocyte images will be acquired from VFN and from cooperating IVF centres (Gynem, s.r.o., Repromeda, s.r.o.). The sequences will be stored and paired with outcome (ploidy status, pregnancy) and also with previously acquired oocyte images. BIOCEV (Academy of sciences of the Czech Republic) will evaluate sperm parameters with respect to oocyte fertilization rate and early embryonic development.

ELIGIBILITY:
Inclusion Criteria:

* Intracytoplasmatic Sperm Injection
* Preimplantation genetic testing
* Time lapse embryo record
* Singned informed consent

Exclusion Criteria:

* Gynecological diseases
* Genetical diseases of parents

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertility couples, where ICSI and PDT are indicated
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
The relative number of embryos whose ploidy was correctly predicted by AI | 1 hour
  Using an AI based non-invasive method of selecting a high-quality and genetically healthy embryos will undoubtably improve clinical and diagnostic practice and reduce costs in the field of infertility treatment. Both the segmentation and classification training will be based on expert annotations. The approach should lead to a classification accuracy at least 70%.

CONTACTS AND LOCATIONS:
Locations (4):
- Czechia (4):
  - General University Hospital in Prague, Prague
  - Czech Technical University in Prague, Prague
  - Institute of Physics AS CR, Prague
  - Biocev As Cr, Vestec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Loendersloot LL, van Wely M, Limpens J, Bossuyt PM, Repping S, van der Veen F. Predictive factors in in vitro fertilization (IVF): a systematic review and meta-analysis. Hum Reprod Update. 2010 Nov-Dec;16(6):577-89. doi: 10.1093/humupd/dmq015. Epub 2010 Jun 25. PMID 20581128
- [Background] Wu B, Shi J, Zhao W, Lu S, Silva M, Gelety TJ. Understanding reproducibility of human IVF traits to predict next IVF cycle outcome. J Assist Reprod Genet. 2014 Oct;31(10):1323-30. doi: 10.1007/s10815-014-0288-y. Epub 2014 Aug 15. PMID 25119191
- [Background] Hanevik HI, Hessen DO. IVF and human evolution. Hum Reprod Update. 2022 Jun 30;28(4):457-479. doi: 10.1093/humupd/dmac014. PMID 35355060
- [Background] Rienzi L, Ubaldi F, Martinez F, Iacobelli M, Minasi MG, Ferrero S, Tesarik J, Greco E. Relationship between meiotic spindle location with regard to the polar body position and oocyte developmental potential after ICSI. Hum Reprod. 2003 Jun;18(6):1289-93. doi: 10.1093/humrep/deg274. PMID 12773461
- [Background] Innocenti F, Fiorentino G, Cimadomo D, Soscia D, Garagna S, Rienzi L, Ubaldi FM, Zuccotti M; SIERR. Maternal effect factors that contribute to oocytes developmental competence: an update. J Assist Reprod Genet. 2022 Apr;39(4):861-871. doi: 10.1007/s10815-022-02434-y. Epub 2022 Feb 15. PMID 35165782